CLINICAL TRIAL: NCT03964844
Title: Incidence, Clinical Characteristics, Strain Characterization, Treatment and Outcome of Clostridium Difficile Infection (CDI) in Hematologic Patients
Brief Title: Clostridium Difficile Infection (CDI) in Hematologic Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Emilio Bouza, Clinical Professor, Hospital General Universitario Gregorio Marañon
Other Study IDs: MICRO.HGUGM.2017-018
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-06

CONDITIONS: C.Difficile Diarrhea
Keywords: hematologic conditions; recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CASE: Patients who had an episode of diarrhoea caused by C. difficile in an hematological unit (2003-2018)
  Interventions: Other: No intervention
- CONTROL: Patients who have had an episode of diarrhoea not caused by C. difficile in an hematological unit (2003-2018)
  Interventions: Other: No intervention
- PROSPECTIVE COHORT: All patients diagnosed with an hematological/oncological disease or with any immunosuppressive condition, who have a positive detection of toxigenic Clostridium difficile in 2019.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The microbiology department prospectively generates a data base of all episodes of Clostridium difficile infection (CDI) in the institution, the investigators will analyse the evolution of the episodes and the incidence per 10,000 days of stay of cases of diagnosed CDI in the Hematological wards and the rest of the hospital during the 2006-2018 period. The investigators will also compare the impact on haematological paediatric population.

In order to analyse the clinical and epidemiological characteristics of CDI in this population, a case and control study will be conducted, reviewing the medical records of patients who have had an episode of diarrhoea caused by C. difficile in an hematological unit, which will be compared with non-hematological patients who have had an CDI episode These patients will be selected randomly from the Microbiology Department database. The sample size will be 400 patients, 200 per arm. The histories will be reviewed according to a pre-established clinical protocol including epidemiological, clinical, therapeutic and evolution variables.

A prospective study in 2019-2020 will also be conducted. The investigators will include all patients diagnosed with an hematological/oncological disease or with any immunosuppressive condition, who have a positive detection of toxigenic Clostridium difficile. Patients will be followed for at least 2 months. For each patient a protocol data will be filled prospectively.

DETAILED DESCRIPTION:
A retrospective case control study (2006-2018) and a prospective study 2019-2020.

Study subjects

All patients diagnosed with a hematological disease who had a detection of toxigenic Clostridium difficile in the laboratory within the 2006-2018 period will be included in the study. Hematological patients with a negative Clostridium difficile infection (CDI) test in the same period will be included as controls, For controls, out of the number of cases within that study period, 200 will be randomly selected with the aid of the Excel software, with the tools randomization (RAND) and INDEX to ensure there is no bias. For each patient a protocol data will be filled retrospectively including the variables listed below.

Additionally, a prospective study in 2019-2020 will also be conducted. We will include all patients diagnosed with an hematological/oncological disease or with any immunosuppressive condition, who have a positive detection of toxigenic Clostridium difficile. Patients will be followed for at least 2 months. For each patient a protocol data will be filled prospectively including the variables listed below.

For all the study period 2006-2018 a total of approximately 200 patients will be included.

For the prospective study 2019-2020 approximately 50 patients will be included.Data collection

For the last 15 years, the institution has kept a prospective record of all episodes of CDI diagnosed in the hospital. This record enables the investigators to assess incidence, incidence density.

The data collected will include age, sex, hospital department or outpatient clinic diagnosis of CDI. Data regarding the underlying conditions and comorbidity factors, clinical data regarding the CDI episode days of diarrhea, presence of abdominal pain, abdominal distention, fever, hypotension, toxic megacolon, pseudomembranous colitis, and severity of the CDI episode according to the European Society of Clinical Microbiology and Infectious Diseases (ESCMID) criteria. Analytical data on the day of diagnosis will be recorded. Treatment data will be recorded. Outcome will also recorded be recorded: need for intensive care unit (ICU) admission, need for surgery for CDI episode, recurrence, mortality, and CDI-associated mortality (For more details please find attached the clinical protocol).

The investigators will also assess all the changes regarding different procedures, management and treatments that have occurred during the study period, including all changes in the diagnostic procedures.

From January 2003 to February 2011, diagnosis of CDI was performed on all stool specimens for which a clinical request for C. difficile testing was made. From March 2011 to current days, diagnosis of CDI was also performed in all unformed stool specimens regardless of clinical request.

Laboratory procedure All C. difficile strains will be characterized at molecular level including ribotype, as it is the most widespread method for the molecular typing of Clostridium difficile. It is based on the detection of polymorphisms located in the intergenic region between genes 16S and 23S RNA by polymerase chain reaction (PCR) and electrophoresis on high resolution agarose gels and will be performed according to the technique described by Stubss et al.[13]The resulting ribotyping profiles will be compared to those of international libraries. Additionally antimicrobial susceptibility testing will be performed on these strains.

All analyses will be performed using SPSS 18.0 (SPSS Inc, Chicago, Illinois, USA). Qualitative variables will appear with their frequency distribution. Quantitative variables will be expressed as the median and interquartile range (IQR). Groups will be compared using the Fisher exact test for categorical variables and the t test or Mann-Whitney test for continuous variables. A multivariate logistic regression model will be used to assess predictors of poor outcome of CDI. The odds ratio (OR) and 95% confidence interval (CI) were calculated. A p value <0.05 will be considered significant.

Based on data from our center, for the retrospective part of the study, the total number of hematological patients with CDI corresponding to the study period is approximately 200 patients, all of them will be studied, the sample size for controls will be of 200 patients (ratio 1:1).

For the prospective study, also based in data from our center, approximately 50 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with a hematological disease who had a detection of toxigenic Clostridium difficile in the laboratory within the 2006-2018 period will be included in the study. Hematological patients with a negative CDI test in the same period will be included as controls.
* All patients diagnosed with an hematological/oncological disease or with any immunosuppressive condition, who have a positive detection of toxigenic Clostridium difficile in 2019.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Based on data from our center, for the retrospective part of the study, the total number of hematological patients with CDI corresponding to the study period is approximately 200 patients, all of them will be studied, the sample size for controls will be of 200 patients (ratio 1:1).
  For the prospective study, also based in data from our center, approximately 50 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence | 2006-2020
  number of CDI cases/ 10,000 patient days

SECONDARY OUTCOMES:
Recurrence of CDI | 2006-2020
  The percentage of recurrent CDI episodes with respect of the total number of CDI cases
Mortality attributable to CDI | 2006-2020
  Percentage of patients with CDI whose death is attributed to CDI

CONTACTS AND LOCATIONS:
Overall Officials: Elena Reigadas, PharmD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- HGU Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided